CLINICAL TRIAL: NCT05645419
Title: Development of Chronoprognosis of Myocardial Infarction in Patients With Type 2 Diabetes Mellitus and Development of Personalized Chronoprevention
Brief Title: Chronoprognosis of Myocardial Infarction in Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Center, Kazakhstan (Other)
Responsible Party: Principal Investigator, Kuat Oshakbayev, a principal investigator, University Medical Center, Kazakhstan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AP19675001
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Clinical Study
Keywords: type 2 diabetes mellitus; myocardial infarction; internal personalized biorhythms; external transit rhythms; personalized chronoprevention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- personalized chronoprevention (Experimental): the main group (n=30), where patients with T2D, in addition to their traditional prescriptions, will receive the intervention method of personalized chronoprevention
  Interventions: Behavioral: personalized chronoprevention
- traditional prescriptions (No Intervention): the control group (n=30), where patients with T2D will only be under observation in addition to their traditional prescriptions

INTERVENTIONS:
Behavioral: personalized chronoprevention — Chronobiological variables: dynamic and static position of the planets of the solar system, moon, sun, constellations; angles/degrees of celestial objects above/below the horizon; angular interactions between celestial objects; the moment/time of the patients' birth; moment/time of MI occurrence; latitude / longitude of the place of birth of the patients, as well as the occurrence of MI (event); the degree of influence of celestial objects in relation to the constellations, where they were at a particular personal event / points of the patient.
  Arms: personalized chronoprevention

SUMMARY:
Purpose: To develop a mathematical model for the occurrence of MI in patients with T2D by studying the relationship between the internal personalized biorhythms of the patients and the external transit rhythms of space objects; to develop and implement a personalized method of chrono-prevention of MI in patients with T2D.

Obejectives:

1.1 To investigate patterns of the influence of external transit rhythms of space objects on the occurrence of MI in patients with T2D: an observational study using clinical databases.

1.2 To investigate patterns of influence of cyclic activity of helio- and geophysical phenomena in the interplanetary medium on the occurrence of MI in patients with T2D.

2. Develop a mathematical model for predicting the occurrence of MI in patients with T2D, based on the identification of the relationship patterns between the internal personalized biorhythms of these patients and the external transit rhythms of space objects.

3. To investigate the effectiveness of the mathematical model for predicting the occurrence of MI in patients with T2D for the purpose of personalized chrono-prevention: a randomized clinical trial.

DETAILED DESCRIPTION:
Participants and study design.

1. Study of the influence of external transit rhythms of space objects, as well as the cyclic activity of helio- and geophysical phenomena in the interplanetary medium on the occurrence of MI in patients with T2D combining population based and clinical data.

   For a retrospective population study, all patients aged 30-65 years with T2D (MI+/-) from the republican database of the Ministry of Health of the Republic of Kazakhstan (MoH) over the past 10 years will be included.

   For a prospective population trial ≥150 patients aged 30-65 years with T2D (MI+/-) will be included.
2. Mathematical and statistical analysis of the collected chrono-geo-biological and clinical data and data on the relationship between the internal personalized biorhythms of the patients and the external transit rhythms of space objects with the definition of "critical periods" as well as the cyclic activity of helio- and geophysical phenomena in the interplanetary medium. Study duration: 12-24 weeks.
3. Study of the effectiveness of the developed mathematical model for predicting the occurrence of MI in patients with T2D in a pilot prospective randomized clinical trial (personalized chronoprophylaxis). The study will include at least 60 patients aged 30-65 years of both sexes with moderate T2D: 1) the main group (n≥30), where patients with T2D will additionally receive personalized chronoprevention intervention; 2) the control group (n≥30), where patients with T2D will only be under observation.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 30-65 years of both sexes
* severe-to-moderate subcompensated stage of T2D without MI
* decompensated stage of T2D without MI

Exclusion Criteria:

* compensated stage of T2D without MI
* patients with T2D and with MI

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with myocardial infarction | 24 weeks
  occurence of myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Altay N Nabiyev, Dr., Study Director — University Medical Center, Kazakhstan
Locations (1):
- Kuat Pernekulovich Oshakbayev, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: Yes
we will make our data available to any investigator/reviewer on their own request, so that the personal privacy of our patients cannot be compromised.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: data will become available to the end of 2025 year, and for 3 years
Access Criteria: by requesting